CLINICAL TRIAL: NCT03340870
Title: Pharmacokinetics of Sonazoid™ Following Intravenous Bolus Injection in Healthy Volunteers
Brief Title: A Study to Evaluate Pharmacokinetics of Sonazoid™ Following Intravenous Bolus Injection in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GE-045-001; GE-045-001 (Other: GE HealthCare)
Record Dates: First submitted 2017-11-02; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Healthy
MeSH Terms: interventions — Sonazoid; perfluorobutane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sonazoid™ 0.12 microliter (µl) (Experimental): Participants will receive single intravenous (I.V) bolus injection of Sonazoid™ 0.12 µl microbubbles (MB)/kilogram (kg) body weight.
  Interventions: Drug: Sonazoid™
- Sonazoid™ 0.60 µl (Experimental): Participants will receive single I.V bolus injection of Sonazoid™ 0.60 µl MB/kg body weight.
  Interventions: Drug: Sonazoid™

INTERVENTIONS:
Drug: Sonazoid™ — Single Dose of Sonazoid™ lipid-stabilised aqueous suspension of perfluorobutane (PFB) gas microbubbles.
  Other Names: perfluorobutane

SUMMARY:
The primary purpose of this study is to determine the Pharmacokinetics (PK) data of perfluorobutane (PFB) in blood and exhaled air following intravenous (I.V.) bolus injection of Sonazoid™ in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria: Participants may be included in the study if they meet all of the following criteria:

* Participant is between 18 and 45 years of age
* Participant is male, or a female who was either surgically sterile (has a documented bilateral oophorectomy and/or documented hysterectomy), postmenopausal (cessation of menses for more than 1 year), or non-lactating, or if of childbearing potential the results of a serum or urine human chorionic gonadotropin pregnancy test, performed on the day of Sonazoid™ administration (with the result known before IMP administration), were negative
* Participant is able and willing to comply with study procedures and provide signed and dated informed consent
* Participant has a body mass index of 19 to 26
* Participant has agreed not to smoke from 2 hours before to 5 hours after Sonazoid™ administration
* Participant has agreed to avoid strenuous physical activity from 1 week before Sonazoid™ administration until the end of the study follow-up
* Participant has no history of alcohol or substance abuse, and has agreed to no intake of alcohol or drugs for 48 hours before Sonazoid™ administration and until the end of the study follow-up
* Participant has a normal health status, as judged by medical history and physical examination at screening
* Normal 12-lead electrocardiogram (ECG) at screening. Minor abnormalities considered by the investigator to be of no clinical importance are permitted
* Normal blood and urine clinical chemistry variables at screening. Isolated or minimally out-of-range values considered by the investigator to be of no clinical importance are permitted
* No regular use of concomitant medication, except for routine use of supplemental oestrogen

Exclusion Criteria:

* Participant was previously included in this study
* Participation in another clinical trial with an unregistered medicinal product, or less than 30 days have passed since completing participation in such a trial
* Participant has a history of allergies to eggs or egg products (i.e., manifested by full body rash, respiratory difficulty, oral and laryngeal swelling, hypotension or shock)
* Donation of >500 milliliter (mL) blood in the 12 weeks before Sonazoid™ administration
* Participant with congenital heart defects, including right-to-left, bi-directional, or transient right-to-left cardiac shunts
* Participant has positive test results for hepatitis B, hepatitis C, or human immunodeficiency virus

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10-20 (Actual); Primary Completion 2014-11-20 (Actual); Study Completion 2014-11-20 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Versus Time Curve from Time Zero to the Last Time- Point (AUC 0-last), AUC from Time Zero to Infinity (AUC0-infinity∞) After Single Dose in Blood | Pre dose and at 0.5, 1, 2, 5, 10, 15, 30, 60, 120 minutes and 4 hours post dose
Area Under the Concentration Versus Time Curve from Time Zero to the Last Time- Point (AUC 0-last), AUC from Time Zero to Infinity (AUC0-Infinity∞) After Single Dose in Exhaled Air | Pre dose and at 1, 3, 6, 9, 16, 31, 61, 121 minutes and 4 hours post dose
Percentage of the Extrapolated Area to Total Area (% AUC ext) After Single Dose in Blood | Pre dose and at 0.5, 1, 2, 5, 10, 15, 30, 60, 120 minutes and 4 hours post dose
Percentage of the Extrapolated Area to Total Area (% AUC ext) After Single Dose in Exhaled Air | Pre dose and at 1, 3, 6, 9, 16, 31, 61, 121 minutes and 4 hours post dose
Elimination Rate Constant (kel) in Blood | Pre dose and at 0.5, 1, 2, 5, 10, 15, 30, 60, 120 minutes and 4 hours post dose
Elimination Rate Constant (kel) in Exhaled Air | Pre dose and at 1, 3, 6, 9, 16, 31, 61, 121 minutes and 4 hours post dose
Elimination Half-life (t½) in Blood | Pre dose and at 0.5, 1, 2, 5, 10, 15, 30, 60, 120 minutes and 4 hours post dose
Elimination Half-life (t½) in Exhaled Air | Pre dose and at 1, 3, 6, 9, 16, 31, 61, 121 minutes and 4 hours post dose
Clearance (Cl) in Blood | Pre dose and at 0.5, 1, 2, 5, 10, 15, 30, 60, 120 minutes and 4 hours post dose
Clearance (Cl) in Exhaled Air | Pre dose and at 1, 3, 6, 9, 16, 31, 61, 121 minutes and 4 hours post dose
Maximum Observed Concentration (Cmax) in Blood | Pre dose and at 0.5, 1, 2, 5, 10, 15, 30, 60, 120 minutes and 4 hours post dose
Maximum Observed Concentration (Cmax) in Exhaled Air | Pre dose and at 1, 3, 6, 9, 16, 31, 61, 121 minutes and 4 hours post dose
Time at which Cmax is reached (tmax) in Blood | Pre dose and at 0.5, 1, 2, 5, 10, 15, 30, 60, 120 minutes and 4 hours post dose
Time at which Cmax is reached (tmax) in Exhaled Air | Pre dose and at 1, 3, 6, 9, 16, 31, 61, 121 minutes and 4 hours post dose
Volume of Distribution (Vd) in Blood | Pre dose and at 0.5, 1, 2, 5, 10, 15, 30, 60, 120 minutes and 4 hours post dose
Volume of Distribution (Vd) in Exhaled Air | Pre dose and at 1, 3, 6, 9, 16, 31, 61, 121 minutes and 4 hours post dose

SECONDARY OUTCOMES:
Percentage of Participants With Treatment-Related Adverse Events (AEs) | Up to 72 hours after first administration of investigational medicinal product (IMP)
Percentage of Participants With Abnormal Laboratory Values | Up to 4 hours post dose
Percentage of Participants With Abnormal Vital Signs | Up to 4 hours post dose
Percentage of Participants With Injection Site Reactions | Up to 4 hours post dose
Percentage of Participants With Abnormal Physical Examinations | Up to 4 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Francois Tranquart, MD, PhD, Study Chair — GE Healthcare
Locations (1):
- Beijing Chao-Yang Hospital, Capital Medical University, NO. 8 Gongren Tiyuchang Nanlu, Chaoyang, Beijing Municipality, China